CLINICAL TRIAL: NCT06773143
Title: Effect of Subanesthetic Dose of Esketamine on Sleep Quality in Patients With Breast Cancer After Chemotherapy
Brief Title: Effect of Subanesthetic Dose of Esketamine on Sleep Quality
Acronym: EOSDOEOSQ
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KY20240514-05-KS-01; ZKX21038 (Other Grant/Funding Number: Nanjing Municipal Health Commission)
Record Dates: First submitted 2025-01-01; First posted 2025-01-14 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Insomnia; Breast Cancer Surgery; Esketamine
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- esketamine group (Experimental): After the patient is induced with general anesthesia, esketamine (0.3 mg/kg/h) will be continuously infused during the operation until the end of the operation.
  Interventions: Drug: Esketamine at low dose
- control group (Placebo Comparator): After the patient's general anesthesia induction is completed, normal saline will be continuously infused until the end of the operation, and the infusion volume is the same as that of the esketamine group.
  Interventions: Other: Normal Saline (0.9% NaCl)

INTERVENTIONS:
Drug: Esketamine at low dose — After the induction of general anesthesia, patients in the esketamine group will receive a continuous infusion of esketamine (0.3 mg/kg/h) until the end of the operation.
  Arms: esketamine group
Other: Normal Saline (0.9% NaCl) — After the patient's general anesthesia induction is completed, normal saline will be continuously infused until the end of the operation, and the infusion volume is the same as that of the esketamine group.
  Arms: control group

SUMMARY:
The goal of this clinical trial is to explore whether subanesthetic doses of esketamine can improve the sleep quality of patients undergoing modified radical mastectomy for breast cancer. In this study, 184 people are expected to participate from admission to three days after surgery.

The process requires participants to cooperate with the completion of the digital rating scale, the Athens Insomnia Scale, the Visual Analog Pain Rating Scale, the Hospital Anxiety and Depression Rating Scale, and the collection of venous blood for research indicators (IL-6, TNF-α, cor, BDNF).

If participants agree to participate in this study, the investigators will assign a unique identification number to each participant and create a medical record for participants.

One day before surgery, the investigators will conduct assessments using the Athens Insomnia Scale, the Visual Analog Pain Rating Scale, and the Hospital Anxiety and Depression Scale, and collect approximately 6 mL of venous blood.

One day after surgery, the investigators will repeat the assessments using the Athens Insomnia Scale, the Visual Analog Pain Rating Scale, and the Hospital Anxiety and Depression Scale. Additionally, the investigators will collect another 6 mL of venous blood and monitor the use of analgesics.

The investigators will follow up with participants three days after the surgery. During this follow-up, investigators will assess any sleep disturbances, administer the Hospital Anxiety and Depression Scale, and review the use of analgesics.

DETAILED DESCRIPTION:
In 2020, breast cancer became the most common cancer worldwide. Treatment methods for breast cancer include surgery, chemotherapy, and endocrine therapy, with surgery remaining the primary treatment option. The emergence of neoadjuvant chemotherapy has expanded the indications for breast cancer surgery, providing surgical opportunities for patients with late-stage clinical staging and a strong desire for breast preservation. Neoadjuvant chemotherapy has the effects of reducing tumor size, lowering clinical staging, assessing the tumor's sensitivity to chemotherapy drugs, and inhibiting tumor cell proliferation. However, chemotherapy, while treating the disease, also causes numerous adverse reactions that directly or indirectly lead to sleep disturbances in patients.

Sleep disturbances reduce cognitive function, immune function, and quality of life in breast cancer chemotherapy patients, with an incidence of sleep disturbances during chemotherapy reaching 80%. These patients, when undergoing surgery, are highly prone to postoperative sleep disturbances (Postoperative Sleep Disturbance, PSD) due to factors such as preoperative sleep disturbances, fear and anxiety about surgery, inflammatory responses, and pain. This negatively impacts their recovery process.

PSD refers to changes in sleep structure and quality in the early postoperative period. It is a clinical syndrome characterized by disturbances in the sleep-wake rhythm following surgery, leading to abnormal sleep quality or sleep behavior, usually manifesting as reduced rapid eye movement (REM) sleep, prolonged wakefulness, and fragmented sleep. There is no unified standard for the duration of PSD, as it varies according to disease type, surgical procedure, and individual differences. Generally, it occurs within a short time after surgery, such as 1-3 days postoperatively. PSD significantly affects the postoperative circadian rhythm, pain levels, inflammatory responses, cognitive function, and cardiovascular outcomes, leading to prolonged recovery time. Clinically, both pharmacological and non-pharmacological interventions are used, with pharmacological treatments primarily involving benzodiazepines, which increase sleep duration and reduce sleep latency. Studying short-term sleep disturbances helps identify and reduce postoperative complications, such as delirium, infections, and cardiovascular events, thus accelerating recovery, improving patient safety, and promoting multidisciplinary collaboration. However, there is limited research on the preventive improvement of sleep quality.

Esketamine, a non-competitive N-methyl-D-aspartate receptor (NMDA) antagonist, is the right-handed isomer of ketamine. It shares a similar pharmacological mechanism with ketamine, but its potency is higher. The most important effect of esketamine is its ability to inhibit the NMDA receptor-mediated glutamate entry into the GABA nervous system, causing excitability changes in the cortex and limbic system, ultimately leading to loss of consciousness. Sub-anesthetic doses of esketamine (0.5 mg/kg, 40-minute intravenous infusion) have been shown to produce rapid and sustained antidepressant effects in patients with treatment-resistant major depressive disorder (MDD).

Additionally, intravenous administration of esketamine at 0.2-0.4 mg/kg (single infusion over 40 minutes) has demonstrated rapid and potent antidepressant effects in the treatment of refractory depression. Apart from its antidepressant effects, esketamine has been proven to improve sleep disturbances in patients with MDD and sleep issues, suggesting that esketamine has potential as a treatment for sleep disorders. Some studies indicate that the antidepressant effect of esketamine is related to the neurobiological structure of wakefulness, sleep, and circadian rhythms. Animal studies also suggest that esketamine can modulate the NF-κB signaling pathway and oxidative stress, inhibiting the release of downstream inflammatory factors, thereby reducing surgical-induced inflammatory damage and playing an anti-anxiety, antidepressant role to improve postoperative recovery quality. However, it remains unclear whether continuous low-dose infusion of esketamine during surgery can reduce the incidence of PSD. This study aims to investigate the impact of continuous infusion of esketamine during surgery on postoperative sleep quality in patients undergoing modified radical mastectomy for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with breast cancer by pathology and immunohistochemistry
2. Patients receiving neoadjuvant chemotherapy
3. Age 18 to 65 years old; d) ;
4. ASA grade Ⅰ - Ⅲ
5. BMI 18 to 30 kg/m2

Exclusion Criteria:

* 1: Patients refuse to participate in the study

  2: BMI > 30 kg/m2

  3: Recent history of drug abuse

  4: Allergy to or contraindications to esketamine

  5: Cognitive dysfunction or inability to communicate

  6: Severe dysfunction of important organs such as liver and kidney function

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of PSD on postoperative day -1 | the first day after surgery
  On the first day after surgery, NRS ≥ 6 or AIS ≥ 6.PSD is defined as a numeric rating scale (NRS) ≥6 or Athens Insomnia Scale (AIS) ≥6, indicating that sleep is repeatedly disturbed or worse throughout the night. NRS scores range from 0 to 10, with 0 representing excellent or good sleep and 10 representing inability to sleep all night. AIS consists of 8 items: nighttime awakenings, sleep induction, final awakening, total sleep time, sleep quality, well-being, functional ability, and daytime sleepiness.

SECONDARY OUTCOMES:
static Visual Analog Scale score on postoperative day -2 | on postoperative day -2
  The painful visual simulation table of pain is a tool for evaluating the strength of pain. It is usually composed of a 10 -centimeter straight line. The two ends are marked as "painless" and "most pain". Patients are marked on the straight line according to their degree of pain.
dynamic Visual Analog Scale score on postoperative day -2 | on postoperative day -2
  The painful visual simulation table of pain is a tool for evaluating the strength of pain. It is usually composed of a 10 -centimeter straight line. The two ends are marked as "painless" and "most pain". Patients are marked on the straight line according to their degree of pain.
anxiety and depression score on the day before surgery | the day before surgery
  The hosp Anxiety and depression scale is a self-evaluation table commonly used in evaluation of anxiety and depression . It contains 14 problems, divided into two sub-meters, and each sub-meter contains 7 items: Anxious sub -meter: Evaluate the anxiety experience of patients in the past week. Depression Meter: Evaluate the depression experience of patients in the past week. Each problem has four levels of options, corresponding to different scores, usually 0 to 3 points. The scoring standard is as follows: 0-7 points: normal 8-10 points: may be mild depression/anxiety
The incidence of PSD on postoperative day -3 | he third day after surgery
  On the third day after surgery, NRS ≥ 6 or AIS ≥6.
The incidence of PSD on postoperative day -5 | On the fifth day after surgery
  On the fifth day after surgery, NRS ≥ 6 or AIS ≥6.
The incidence of PSD on postoperative day 7 | On the seventh day after surgery
  On the seventh day after surgery, NRS ≥ 6 or AIS ≥6.
static Visual Analog Scale score on postoperative day -1 | on postoperative day -1
  The painful visual simulation table of pain is a tool for evaluating the strength of pain. It is usually composed of a 10 -centimeter straight line. The two ends are marked as "painless" and "most pain". Patients are marked on the straight line according to their degree of pain.
dynamic Visual Analog Scale score on postoperative day -1 | on postoperative day -1
  The painful visual simulation table of pain is a tool for evaluating the strength of pain. It is usually composed of a 10 -centimeter straight line. The two ends are marked as "painless" and "most pain". Patients are marked on the straight line according to their degree of pain.
BDNF on postoperative day -1 | on postoperative day -1
TNFα on postoperative day -1 | on postoperative day -1
IL-6 on postoperative day -1 | on postoperative day -1

OTHER OUTCOMES:
IL-6 blood on the day before surgery | the day before surgery
TNFα on the day before surgery | the day before surgery
BDNF on the day before surgery | the day before surgery

CONTACTS AND LOCATIONS:
Overall Officials: xiaoliang wang, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
Due to the relevant regulations of our hospital and considering the personal privacy of patients, we will not provide IPD. However, if necessary, you can also contact the researcher in charge of this study to view the relevant data to prove the authenticity of this study.

REFERENCES:
- [Background] Sun J, Wang XD, Liu H, Xu JG. Ketamine suppresses endotoxin-induced NF-kappaB activation and cytokines production in the intestine. Acta Anaesthesiol Scand. 2004 Mar;48(3):317-21. doi: 10.1111/j.0001-5172.2004.0312.x. PMID 14982564
- [Background] Kohtala S, Alitalo O, Rosenholm M, Rozov S, Rantamaki T. Time is of the essence: Coupling sleep-wake and circadian neurobiology to the antidepressant effects of ketamine. Pharmacol Ther. 2021 May;221:107741. doi: 10.1016/j.pharmthera.2020.107741. Epub 2020 Nov 12. PMID 33189715
- [Background] Song B, Zhu J. A Novel Application of Ketamine for Improving Perioperative Sleep Disturbances. Nat Sci Sleep. 2021 Dec 25;13:2251-2266. doi: 10.2147/NSS.S341161. eCollection 2021. PMID 34992482
- [Background] Song B, Zhu JC. Mechanisms of the Rapid Effects of Ketamine on Depression and Sleep Disturbances: A Narrative Review. Front Pharmacol. 2021 Dec 14;12:782457. doi: 10.3389/fphar.2021.782457. eCollection 2021. PMID 34970147
- [Background] Wang M, Zhang B, Zhou Y, Wang C, Zheng W, Liu W, Zhan Y, Lan X, Ning Y. Sleep improvement is associated with the antidepressant efficacy of repeated-dose ketamine and serum BDNF levels: a post-hoc analysis. Pharmacol Rep. 2021 Apr;73(2):594-603. doi: 10.1007/s43440-020-00203-1. Epub 2021 Jan 2. PMID 33387333
- [Background] Bahji A, Vazquez GH, Zarate CA Jr. Comparative efficacy of racemic ketamine and esketamine for depression: A systematic review and meta-analysis. J Affect Disord. 2021 Jan 1;278:542-555. doi: 10.1016/j.jad.2020.09.071. Epub 2020 Sep 23. PMID 33022440
- [Background] Murrough JW, Iosifescu DV, Chang LC, Al Jurdi RK, Green CE, Perez AM, Iqbal S, Pillemer S, Foulkes A, Shah A, Charney DS, Mathew SJ. Antidepressant efficacy of ketamine in treatment-resistant major depression: a two-site randomized controlled trial. Am J Psychiatry. 2013 Oct;170(10):1134-42. doi: 10.1176/appi.ajp.2013.13030392. PMID 23982301
- [Background] Luo M, Song B, Zhu J. Sleep Disturbances After General Anesthesia: Current Perspectives. Front Neurol. 2020 Jul 8;11:629. doi: 10.3389/fneur.2020.00629. eCollection 2020. PMID 32733363
- [Background] Qiu D, Wang XM, Yang JJ, Chen S, Yue CB, Hashimoto K, Yang JJ. Effect of Intraoperative Esketamine Infusion on Postoperative Sleep Disturbance After Gynecological Laparoscopy: A Randomized Clinical Trial. JAMA Netw Open. 2022 Dec 1;5(12):e2244514. doi: 10.1001/jamanetworkopen.2022.44514. PMID 36454569
- [Background] Matthews EE, Berger AM, Schmiege SJ, Cook PF, McCarthy MS, Moore CM, Aloia MS. Cognitive behavioral therapy for insomnia outcomes in women after primary breast cancer treatment: a randomized, controlled trial. Oncol Nurs Forum. 2014 May;41(3):241-53. doi: 10.1188/14.ONF.41-03AP. PMID 24650832